CLINICAL TRIAL: NCT01199939
Title: A Multicenter, Single Arm, Open-Label Study of the Once Daily Combination of Etravirine and Darunavir/Ritonavir As Dual Therapy in Early Treatment-Experienced Patients
Brief Title: A Study of the Once Daily Combination of Etravirine and Darunavir/Ritonavir As Dual Therapy in Early Treatment-Experienced Patients
Acronym: INROADS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec, Inc (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017149; TMC125HIV4007 (Other: Tibotec, Inc.)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-10

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Human Immunodeficiency Virus; HIV; Etravirine; Darunavir; Prezista; Intelence; Ritonavir; INROADS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — etravirine; Ritonavir; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ETR + DRV/rtv (Experimental): Darunavir 800mg once daily orally for 48 weeks,Etravirine 400mg once daily orally for 48 weeks,Ritonavir 100mg once daily orally for 48 weeks
  Interventions: Drug: Etravirine; Drug: Ritonavir; Drug: Darunavir

INTERVENTIONS:
Drug: Etravirine — 400mg once daily orally for 48 weeks
Drug: Ritonavir — 100mg once daily orally for 48 weeks
Drug: Darunavir — 800mg once daily orally for 48 weeks

SUMMARY:
This study is a Phase II single arm, open-label, multicenter, study of 50 human immunodeficiency virus-1 (HIV) infected adult patients, all of whom will receive etravirine (ETR) 400mg and DRV/r 800/100mg each given orally once daily. This trial is designed to evaluate the efficacy of the aforementioned ARV regimen, as measured by the percentage of patients with HIV RNA <50 copies/mL at 48 weeks, in early treatment-experienced HIV-infected patients. In addition to general safety parameter measurements, this trial will also assess changes in metabolic, inflammatory, immune restoration, and bone markers. Screening will occur over a 6-week period. The primary endpoint will be assessed at Week 48, and the treatment period is 48 weeks. The end of study endpoint will be met by either completing the Week 48 visit, or by early termination from the study for any reason.

DETAILED DESCRIPTION:
This study is a Phase II single arm, open-label, multicenter, (all people involved know the identity of the intervention) study of 50 HIV-1 infected adult patients, all of whom will receive ETR 400mg and darunavir (DRV)/r 800/100mg each given orally once daily. This trial is designed to evaluate the efficacy of the aforementioned ARV regimen, as measured by the percentage of patients with HIV ribonucleic acid (RNA) <50 copies/mL at 48 weeks, in early treatment-experienced HIV-infected patients. In addition to general safety parameter measurements, this trial will also assess changes in metabolic, inflammatory, immune restoration, and bone markers. Screening will occur over a 6-week period. The trial schedule includes a Baseline Visit (Day 1), Open-label Treatment Phase (Weeks 4, 8, 12, 16, 20, 24, 30, 36, 42, 48/ Early Withdrawal) and a Post-treatment Phase (4 Week Follow-Up) visit. In addition, all patients will have two pharmacokinetic (PK) samples drawn at Weeks 4 and 24, A single PK sample will be drawn at Weeks 12, 36, and 48 (or early withdrawal visit). There will also be a substudy conducting 24 hour intensive PK at week 4 for a subset of patients. For patients who consent, genotyping for CYP2C9 and CYP2C19 will be performed at Baseline. A Modified Medication Adherence Self-Report Inventory (M-MASRI) questionnaire will be collected, which is a patient-reported survey to assess adherence to medication taking. The primary endpoint will be assessed at Week 48, and the treatment period is 48 weeks. The end of study endpoint will be met by either completing the Week 48 visit, or by early termination from the study for any reason. ETR 400mg once daily for 48 weeks and DRV 800mg once daily for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18 years or above
* Patients with documented HIV-1 infection
* On current HAART regimen for at least 12 weeks continuous duration at screening, and with an HIV-1 plasma viral load above 500 HIV-1 RNA copies/mL by site's currently utilized viral load assay (Note: For the purposes of this study, HAART is defined as treatment with a combination of 3 or more HIV antiretroviral medications from at least 2 different classes of medications (NRTIs, NNRTIs, PIs, integrase inhibitors, CCR5 antagonists, fusion inhibitors))
* No more than 2 previous virologic failures while on PI-containing HAART regimens where virologic failure is generally defined as either a lack of suppression of the subjects' viral load to lower limit of quantification (per standard assay historically used in care) after 24 weeks of treatment or, rebound of a previously suppressed viral load (undetectable per investigator's standard of care) to detectable limits and without demonstrated re-suppression on the same regimen
* Demonstrated phenotypic sensitivity to both etravirine and darunavir based on resistance testing at Screening (FC= 2.9 for etravirine and FC = 10.0 for darunavir using the PhenoSense GT)
* The absence of all of the following Resistance Associated Mutations (RAMS) at baseline: For Darunavir: V11I, V32I, L33F, I47V, I50V, I54L/M, T74P, L76V, I84V, L89V
* For Etravirine: L100I, E138A, I167V, V179D, V179F, Y181I, Y181V, G190S
* 7. CD4 count = 50 cells/mm3.

Exclusion Criteria:

* Primary HIV-1 infection
* Previously documented HIV-2 infection
* Use of disallowed concomitant therapy

Any condition (including but not limited to alcohol and drug use), which, in the opinion of the investigator, could compromise the patient's safety or adherence to the protocol

* Life expectancy less than 6 months according to the judgment of the investigator
* Patient has any currently active AIDS defining illness (Category C conditions according to the Center for Disease Control [CDC] Classification System for HIV infection 1993
* with the following exceptions, which must be discussed with the sponsor prior to enrollment: Stable cutaneous Kaposi's Sarcoma (i.e., no pulmonary or gastrointestinal involvement other than oral lesions) that is unlikely to require any form of systemic therapy during the trial period
* Wasting syndrome due to HIV infection if, in the investigator's opinion, it is not actively progressive and its treatment does not require hospitalization or compromise the patient's safety or compliance to adhere to trial-related procedures. If the patient is on maintenance therapy (which may include Growth Hormone, appetite stimulants and anabolic steroids) for previously diagnosed wasting syndrome, he/she may be eligible for the trial. Note: An AIDS defining illness not clinically stabilized for at least 30 days will be considered clinically active. Note: Primary and secondary prophylaxis for an AIDS defining illness is allowed in case the medication used is not part of the disallowed medications
* Any active clinically significant disease (e.g., pancreatitis, cardiac dysfunction) or findings during screening of medical history, laboratory or physical examination that, in the investigator's opinion, would compromise the patient's safety or the outcome of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec, Inc. Clinical Trial, Study Director — Tibotec, Inc
Locations (23):
- United States (22):
  - Long Beach, California
  - Los Angeles, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Ft. Pierce, Florida
  - Miami, Florida
  - Orlando, Florida
  - Decatur, Georgia
  - Macon, Georgia
  - Berkley, Michigan
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Neptune City, New Jersey
  - Buffalo, New York
  - Manhasset, New York
  - Charlotte, North Carolina
  - Austin, Texas
  - Dallas, Texas
  - Harlingen, Texas
  - Houston, Texas
  - Seattle, Washington
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Ruane PJ, Brinson C, Ramgopal M, Ryan R, Coate B, Cho M, Kakuda TN, Anderson D; INROADS study investigators. The Intelence aNd pRezista Once A Day Study (INROADS): a multicentre, single-arm, open-label study of etravirine and darunavir/ritonavir as dual therapy in HIV-1-infected early treatment-experienced subjects. HIV Med. 2015 May;16(5):288-96. doi: 10.1111/hiv.12211. Epub 2015 Jan 14. PMID 25585528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 29 March 2010 and 5 October 2012 and recruited patients from US (17 sites) and Puerto Rico (1 site).
Pre-assignment Details: 54 participants were treated with Etravirine and Darunavir/ritonavir in this study.
Groups:
- ETR + DRV/Rtv: Etravirine (ETR) 400mg + Darunavir (DRV) 800mg/Ritonavir (rtv) 100mg once daily orally for 48 weeks
Period: Overall Study
Arm/Group | ETR + DRV/Rtv
Started | 54 (Number of enrolled participants)
Completed | 41
Not Completed | 13
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 2
Not completed — Reached a virologic endpoint | 4

BASELINE CHARACTERISTICS:
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 42
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 4
  USA | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Virologic Response (CVR) at Week 48
Description: CVR is defined as confirmed plasma Viral Load of less than 50 human immunodeficiency virus - type 1 (HIV-1) ribonucleic acid (RNA) copies/mL.
Time Frame: Week 48
Population: Intent-To-Treat Non-Virologic failure (VF) censored: Participants who took at least one dose of any of the study medications and did not withdraw for reasons other than VF or experienced VF prior to discontinuation. Participants with evaluable data at Week 48
Measure: Number; unit: Participants
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 45
Participants | 40

2. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 4
Time Frame: Baseline (Day 1) and Week 4
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 4
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 52
log10 Copies/mL | -1.77 [-3.2 to 3.1]

3. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 8
Time Frame: Baseline (Day 1) and Week 8
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 8
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 50
log10 Copies/mL | -2.04 [-3.3 to -0.5]

4. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 12
Time Frame: Baseline (Day 1) and Week 12
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 12
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 45
log10 Copies/mL | -2.18 [-3.6 to -0.1]

5. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 16
Time Frame: Baseline (Day 1) and Week 16
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 16
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 45
log10 Copies/mL | -2.29 [-4.0 to -0.5]

6. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 20
Time Frame: Baseline (Day 1) and Week 20
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 20
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 44
log10 Copies/mL | -2.27 [-4.0 to -0.5]

7. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 24
Time Frame: Baseline (Day 1) and Week 24
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 24
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 45
log10 Copies/mL | -2.17 [-3.9 to -0.2]

8. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 30
Time Frame: Baseline (Day 1) and Week 30
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 30
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 43
log10 Copies/mL | -2.28 [-4.0 to -0.5]

9. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 36
Time Frame: Baseline (Day 1) and Week 36
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 36
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 42
log10 Copies/mL | -2.24 [-3.9 to -0.5]

10. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 42
Time Frame: Baseline (Day 1) and Week 42
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 42
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 41
log10 Copies/mL | -2.29 [-3.9 to -0.5]

11. Secondary Outcome: Change From Baseline in Log10 Plasma Human Immunodeficiency Virus - Type 1 (HIV-1) Viral Load at Week 48
Time Frame: Baseline (Day 1) and Week 48
Population: Intent-to-treat participants who received at least one dose of any of the study medication with evaluable data at Week 48
Measure: Median (Full Range); unit: log10 Copies/mL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 39
log10 Copies/mL | -2.29 [-3.9 to 2.4]

12. Secondary Outcome: Time to Reach First Confirmed Virologic Response
Description: as for outcome 1
Time Frame: Baseline (Day 1) to Week 48
Population: Intent-To-Treat participants enrolled in the study who took at least one dose of any of the study medications
Measure: Mean (Standard Error); unit: Days
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 54
Days | 82.98 (6.684)

13. Secondary Outcome: Number of Participants With Virologic Failure
Description: Virologic Failure is defined as participant who is a rebounder or a non-responder. Rebounder participant is defined as a participant who is still in the study at Week 12 and first achieves 2 consecutive virologic responses (<50 copies/mL) followed by 2 consecutive non-responses or a discontinued participant (any reason) for which the last observed time point shows a non-response. Non responder participant is defined as a participant who is still in the study at Week 12 and never achieves 2 consecutive responses.
Time Frame: Baseline (Day 1) to Week 48
Population: Intent-To-Treat participants enrolled in the study who took at least one dose of any of the study medications
Measure: Number; unit: Participants
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 54
Participants | 7 (6.684)

14. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) and Cluster of Differentiation 8 (CD8+) Cell Counts at Week 48
Time Frame: Baseline (Day 1) and Week 48
Population: Intent-To-Treat participants enrolled in the study who took at least one dose of any of the study medications
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | ETR + DRV/Rtv
Number analyzed (Participants) | 54
cells/uL
  CD4 | 168 (153.3)
  CD8 | -69 (289.4)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | ETR + DRV/Rtv
Serious Adverse Events (participants affected / at risk) | 3/54
Other Adverse Events (participants affected / at risk) | 28/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETR + DRV/Rtv (N=54)
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Abscess Jaw (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETR + DRV/Rtv (N=54)
Abdominal Pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Sinusitis (Infections and infestations) | 3
Upper Respiratory Tract Infection (Infections and infestations) | 6
Fibrin D Dimer Increased (Investigations) | 3
Low Density Lipoprotein Increased (Investigations) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days